CLINICAL TRIAL: NCT06461429
Title: Platform for Adaptive Trials in Perinatal Units (Core Protocol)
Brief Title: PLatform for Adaptive Trials In Perinatal UnitS - [Core Protocol]
Acronym: PLATIPUS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Melbourne (Other)
Collaborators: University of Auckland, New Zealand (Other); Monash University (Other); The University of Western Australia (Other); La Trobe University (Other); The University of New South Wales (Other); University of Tasmania (Other); Menzies School of Health Research (Other); University of Adelaide (Other); University of Sydney (Other); Mater Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P-CORE-01
Record Dates: First submitted 2024-05-02; First posted 2024-06-17 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2024-06

CONDITIONS: Preterm Birth
Keywords: Preterm infant; Pregnancy; Neonatal complications; Preterm labor
MeSH Terms: conditions — Premature Birth; Obstetric Labor, Premature | interventions — Erythromycin; Amoxicillin; Azithromycin; caffeine citrate

STUDY DESIGN:
Intervention Model Description: PLATIPUS is an Adaptive Platform Trial. Multiple interventions will be tested in this adaptive platform trial and each will be described in domain-specific platform appendices. Pregnant women and people at risk of preterm birth will participate in 'Pregnancy Domains'. Infants born preterm will participate in 'Neonatal Domains'.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The default position is that domains run on the PLATIPUS platform will be randomisation provided on a blinded basis. Blinding, however, may not always be feasible for some interventions and this will be specified in the related Domain-Specific protocol.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pregnancy Domain 01 - PROMOAT: Preterm Rupture Of Membranes Optimal Antibiotics Trial (Experimental): ClinicalTrial.gov Trial Registration: NCT06906757.
  Population: Pregnant women and people with PPROM <37 weeks' gestation and active neonatal management anticipated.
  Interventions: Randomised to receive routinely used broad-spectrum antibiotic prophylaxis
  Interventions: Drug: Erythromycin; Drug: Amoxicillin and Erythromycin; Drug: Azithromycin
- Neonatal Domain 01 - BabyCCINO: Caffeine Citrate to Improve Neonatal Outcomes (Experimental): ClinicalTrial.gov Trial Registration: NCT06972849.
  Population: Very preterm infants born <32 weeks' gestation, up to 10 days old, with any clinical indication to commence caffeine treatment (any of: prevention of apnoea, treatment of apnoea, or with the aim of improving longer-term outcomes.
  Interventions: Randomised to receive high, medium and low-dose caffeine citrate.
  Interventions: Drug: Caffeine citrate 20 mg/kg load and 10 mg/kg daily maintenance.; Drug: Caffeine citrate 30 mg/kg load and 15 mg/kg daily maintenance.; Drug: Caffeine citrate 40 mg/kg load and 20 mg/kg daily maintenance

INTERVENTIONS:
Drug: Erythromycin — Antibiotic. Standard of care. Antibiotics will be administered for 7 days or until delivery (whichever is sooner).
  Arms: Pregnancy Domain 01 - PROMOAT: Preterm Rupture Of Membranes Optimal Antibiotics Trial
Drug: Amoxicillin and Erythromycin — Antibiotic. Antibiotics will be administered for 7 days or until delivery (whichever is sooner).
  Other Names: Amoxycillin
  Arms: Pregnancy Domain 01 - PROMOAT: Preterm Rupture Of Membranes Optimal Antibiotics Trial
Drug: Azithromycin — Antibiotic. Antibiotics will be administered for 7 days or until delivery (whichever is sooner).
  Arms: Pregnancy Domain 01 - PROMOAT: Preterm Rupture Of Membranes Optimal Antibiotics Trial
Drug: Caffeine citrate 20 mg/kg load and 10 mg/kg daily maintenance. — Lower dose caffeine: 20mg/kg load and 10mg/kg/day maintenance. Standard of care. Caffeine will be administered until at least 34+0 weeks' post-menstrual age, with the aim to cease caffeine by 36+0 weeks' post-menstrual age. Caffeine use beyond 36+0 weeks' post-menstrual age will be open-label.
  Arms: Neonatal Domain 01 - BabyCCINO: Caffeine Citrate to Improve Neonatal Outcomes
Drug: Caffeine citrate 30 mg/kg load and 15 mg/kg daily maintenance. — Medium dose caffeine: 30mg/kg load and 15 mg/kg/day maintenance. Caffeine will be administered until at least 34+0 weeks' post-menstrual age, with the aim to cease caffeine by 36+0 weeks' post-menstrual age. Caffeine use beyond 36+0 weeks' post-menstrual age will be open-label.
  Arms: Neonatal Domain 01 - BabyCCINO: Caffeine Citrate to Improve Neonatal Outcomes
Drug: Caffeine citrate 40 mg/kg load and 20 mg/kg daily maintenance — Higher dose caffeine: 40mg/kg load and 20mg/kg/day maintenance. Caffeine will be administered until at least 34+0 weeks' post-menstrual age, with the aim to cease caffeine by 36+0 weeks' post-menstrual age. Caffeine use beyond 36+0 weeks' post-menstrual age will be open-label.
  Arms: Neonatal Domain 01 - BabyCCINO: Caffeine Citrate to Improve Neonatal Outcomes

SUMMARY:
PLATIPUS is an adaptive platform trial aimed at improving the health of infants born preterm (before 37 weeks' gestation). PLATIPUS will compare how different treatments and care provided to pregnant women and people at risk of preterm birth and infants born preterm affect infant health.

The main questions PLATIPUS aims to answer are:

1. What effect/s do different treatments/care provided to pregnant women and people at risk of preterm birth have on the health of their infants? (Pregnancy domains)
2. What effect/s do different treatments/care given to infants born preterm have on their health ? (Neonatal domains).

This registration record relates to the PLATIPUS Core (or 'master') protocol which provides guidance for the overall running of the trial. Additional appendices will outline the aims, questions, treatments, and activities for each separate research question (domain). Each Domain-Specific Appendix will be registered separately on ClinicalTrials.gov and will link to this record.

DETAILED DESCRIPTION:
PLATIPUS is a multi-domain, multi-centre international adaptive platform trial and innovative approach to perinatal research.

Preterm birth (birth before 37 weeks' gestation) is a global issue. More than 15 million babies (1 in 10) are born preterm each year. Complications of preterm birth are the leading cause of death and disability among children under five years of age. These contribute to increased risk of all-cause mortality and early death from cardiovascular disease, diabetes and chronic lung disease in later life. There is no single cause of, or pathway to, preterm birth. Treatments during pregnancy aim to prevent or treat complications that can lead to preterm birth in pregnant women and people or reduce the impact of prematurity on neonatal outcomes. Treatments in the neonatal period (period shortly after birth) aim to improve survival and reduce potential morbidities in the preterm infant.

PLATIPUS will initially assess interventions given to pregnant women and people during pregnancy (Participant Group 1) and to preterm infants (Participant Group 2) in the first few days of life. Participants will be randomly allocated to all relevant domains for which they are eligible and provide consent. Using a trial-developed Ordinal Outcome Scale, the effect of pregnancy and/or neonatal interventions on neonatal outcome will be assessed at 42 weeks' post-menstrual age OR at primary hospital discharge, whichever occurs earliest. Secondary outcomes will examine the effect of interventions on individual pregnancy and/or neonatal endpoints, and may be domain-specific. All pregnancy domains will include a 'Maternal Outcome Set' to assess maternal health and intervention safety.

In contrast to conventional clinical trials, PLATIPUS has been designed to examine multiple different treatment options at once within the same platform. Both pregnant and neonatal participants will be randomly assigned to different concurrent treatment options, with an initial focus on treatments already considered as part of clinical care. As the trial advances, novel interventions may also be included. Interventions will be evaluated within domains. A domain is defined as a set of interventions that are intended for a specific health problem or specific therapeutic option.

Bayesian adaptive statistical modelling will be used to evaluate treatment efficacy at regular interim adaptive analyses of the pre-specified outcomes for each intervention in each domain. This will allow determination of the effectiveness of interventions once sufficient data has been accrued, rather than when a pre-specified sample size is reached. Adaptive analyses will compute the posterior probabilities of superiority, futility, inferiority, or equivalence for pre-specified comparisons within domains. Each of these potential conclusions will be pre-defined prior to commencing the intervention domain. Decisions about trial results (e.g., concluding superiority or equivalence) will be based on pre-specified threshold values for posterior probability.

All trial procedures are outlined in the "core" protocol described in this registration. Separate domain protocols with information specific to each intervention included in PLATIPUS will be linked to this registration at separate clinicaltrials.gov records:

ELIGIBILITY:
Potential participants with core platform eligibility AND who meet all domain-specific inclusion criteria and none of the domain-specific exclusion criteria for at least one PLATIPUS domain, will be eligible to 'enrol' in the PLATIPUS trial and randomised to all eligible domains, for which consent has been provided.

CORE PLATFORM ELIGIBILITY - PREGNANCY DOMAINS

Inclusion Criteria: Pregnant women and people must fulfil the following inclusion criteria to be eligible to participate in PLATIPUS:

1. Pregnant and at risk of preterm birth
2. Receiving care at a participating site at the time of eligibility assessment.
3. Meets the eligibility criteria for at least one domain.

Exclusion Criteria: Pregnant women and people who meet the following criteria will be excluded from participation in this trial:

1. Circumstances where death (pregnant woman or person/fetal) is deemed to be imminent and inevitable. The treating team may however decide that providing an opportunity for the pregnant woman or person to participate would be in their and/or their fetus/infant's interest. OR
2. Inability to consent, unless a waiver of consent has been deemed appropriate at domain-level.

CORE PLATFORM ELIGIBILITY - NEONATAL DOMAINS

Inclusion Criteria: Preterm infants must fulfil the following criteria to be eligible to participate in PLATIPUS, infants must be:

1. Born preterm (<37 weeks' gestational age)
2. Receiving care at a participating site at the time of eligibility assessment.
3. Meet the eligibility criteria for at least one domain.

Exclusion Criteria: Preterm infants who meet the following criteria will be excluded from participation in this trial:

1. Circumstances where death (neonatal) is deemed to be imminent and inevitable. The treating team may however decide that providing an opportunity for the infant to participate is in the infant's interest. OR
2. Parental/guardian inability to consent, unless a waiver of consent has been deemed appropriate at domain-level.

DOMAIN-SPECIFIC ELIGIBILITY CRITERIA

Potential participants who meet core platform eligibility criteria will be assessed for eligibility to participate in trial domains available at their hospital. Domain-specific eligibility criteria are outlined in the related Domain-Specific Appendices.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100000 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2050-12-31 (Estimated); Study Completion 2050-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants who progress by at least one level higher on the PLATIPUS Ordinal Outcome Scale | At any time prior to 42 weeks' postmenstrual age or first discharge home from hospital (whichever is earlier).
  The PLATIPUS-Ordinal Outcome Scale ranks the most severe core short-term infant health outcome in the specified time frame.
  Levels 1-15: 1= Well, liveborn infant; 2= Neonatal unit admission for <48 hours; 3= Neonatal unit admission for >/= 48 hours; 4= Non-invasive respiratory support for ≥ 4 hours & < 5 days; 5= Non-invasive respiratory support >/= 5 days; 6= Mechanical ventilation via endotracheal tube for ≥ 4 hours & <7 days; 7= Mechanical ventilation via endotracheal tube for >/=7 days; 8= Moderate respiratory morbidity; 9=Necrotising enterocolitis AND/OR Sepsis; 10= Severe Respiratory Morbidity; 11= Major Surgery; 12= Brain Injury; 13= TWO of severe respiratory morbidity OR major surgery OR brain injury; 14= Severe respiratory morbidity & major surgery & brain injury; 15 = Death.

SECONDARY OUTCOMES:
Number of well liveborn infants | At any time prior to 42 weeks' postmenstrual age or first discharge home from hospital (whichever is earlier).
  Well, liveborn infants who have not met the diagnostic criteria for worse scale outcomes.
  The ordinal outcome scale ranks short-term neonatal outcomes associated with longer-term health in ascending severity. An infant is assigned the outcome that is the highest (worst) for which they have met diagnostic criteria at any time prior to 42 weeks PMA or first hospital discharge (whichever is earlier).
Number of infants admitted to the neonatal unit during primary hospital admission for 48 hours or more. | At any time prior to 42 weeks' postmenstrual age or first discharge home from hospital (whichever is earlier).
  Infants admitted to the neonatal unit during primary hospital admission for 48 hours or more.
Number of infants admitted to neonatal unit during primary hospital admission for <48 hours. | At any time prior to 42 weeks' postmenstrual age or first discharge home from hospital (whichever is earlier).
  Infants admitted to any level of neonatal unit during the birth admission, for less than 48 hours.
Number of infants who received non-invasive positive pressure respiratory support for ≥ 4 hours (excluding delivery room) and less than 5 days. | At any time prior to 42 weeks' postmenstrual age or first discharge home from hospital (whichever is earlier).
  Infants who received non-invasive positive pressure respiratory support for ≥ 4 hours (excluding delivery room) and less than 5 days.
Number of infants who received non-invasive positive pressure respiratory support for 5 days or more. | At any time prior to 42 weeks' postmenstrual age or first discharge home from hospital (whichever is earlier).
  Infants who received non-invasive positive pressure respiratory support for 5 days or more.
Number of infants who received mechanical ventilation via endotracheal tube for ≥ 4 hours (excluding delivery room) and <7 days. | At any time prior to 42 weeks' postmenstrual age or first discharge home from hospital (whichever is earlier).
  Infants who received mechanical ventilation via endotracheal tube for ≥ 4 hours (excluding delivery room) and <7 days.
Number of infants who received mechanical ventilation via endotracheal tube for 7 days or more. | At any time prior to 42 weeks' postmenstrual age or first discharge home from hospital (whichever is earlier).
  Infants who received mechanical ventilation via endotracheal tube for 7 days or more.
Number of infants with moderate respiratory morbidity. | At any time prior to 42 weeks' postmenstrual age or first discharge home from hospital (whichever is earlier).
  Infants with a gestational age <37 weeks who received oxygen therapy at 40 weeks' postmenstrual age.
Number of infants with necrotising enterocolitis OR sepsis. | At any time prior to 42 weeks' postmenstrual age or first discharge home from hospital (whichever is earlier).
  A. Infants with necrotising enterocolitis (NEC), defined as one or more of the following:
  * Radiological diagnosis: Clinical history plus imaging consistent with NEC (pneumatosis intestinalis AND/OR portal venous gas AND/OR persistently dilated loop of bowel on serial imaging)
  * Clinical diagnosis: Clinical history plus abdominal wall cellulitis and a palpable abdominal mass
  AND an intention to treat with broad-spectrum antibiotics for 7 days or more
  OR
  B. Infants with Sepsis Organism (bacterial, fungal or viral) isolated in the blood or CSF by culture or PCR AND an intention to treat with antimicrobials/antivirals for 5 days or more.
  NOTE: Exclude if culture is mixed coagulase negative staphylococcus and/or other skin flora contaminant.
Number of infants with severe respiratory morbidity. | At any time prior to 42 weeks' postmenstrual age or first discharge home from hospital (whichever is earlier).
  Infants with severe respiratory morbidity defined as one or more of the following:
  1. Tracheostomy, assessed at 42+0 weeks' PMA
  2. Discharge home on oxygen AND/OR respiratory support, if discharged prior to or on the day of 40+0 weeks' PMA
  3. Born at <37 weeks' GA AND received respiratory support for 12 hours or more on the day of 40+0 weeks PMA.
Number of participants who underwent major surgery. | At any time prior to 42 weeks' postmenstrual age or first discharge home from hospital (whichever is earlier).
  Infants who underwent major surgery, defined as one of the following:
  * Laparotomy /Laparoscopy
  * Thoracotomy/Thoracoscopy (e.g. ligation of a ductus arteriosus, surgery for NEC etc)
  * Craniotomy / Cranioscopy
  Excludes inguinal hernia repair. Note: Tracheostomy and neurosurgical intervention for post-haemorrhagic hydrocephalus are included in other categories.
Number of infants with brain injury. | At any time prior to 42 weeks' postmenstrual age or first discharge home from hospital (whichever is earlier).
  Infants with brain injury may be diagnosed on ultrasound or magnetic resonance imaging where there is clinical suspicion or request, and includes one or more of the following:
  a. Major intraventricular haemorrhage, unilateral or bilateral, defined as i. Papile Grade 3 or 4 AND/OR ii. Moderate-severe periventricular haemorrhagic infarction b. Cystic periventricular leukomalacia, unilateral or bilateral c. Moderate or severe white matter injury on MRI.Other major ischaemic injury such as arterial stroke or hypoxic ischaemic injury d. Post haemorrhagic hydrocephalus requiring drainage. e. Any cerebellar haemorrhage, excluding punctate lesions (<4mm) that occur in the absence of other brain injury as defined above (12 a, b, c, d and e).
Number of infants with TWO of Brain Injury OR Major Surgery OR Severe Respiratory Morbidity, who did not experience any worse scale outcomes. | At any time prior to 42 weeks' postmenstrual age or first discharge home from hospital (whichever is earlier).
  Infants that meet the definition of TWO of Brain Injury OR Major Surgery OR Severe Respiratory Morbidity (as defined in Scale Categories 10, 11 and 12)
Number of infants with Brain injury AND Major surgery AND Severe respiratory morbidity. | At any time prior to 42 weeks' postmenstrual age or first discharge home from hospital (whichever is earlier).
  Infants that meet the definition of Brain Injury AND Major Surgery AND Severe Respiratory Morbidity (as defined in Scale Categories 10, 11 and 12)
Number of infants who died | At any time prior to 42 weeks' postmenstrual age or first hospital discharge home from hospital (whichever is earlier).
  Death includes fetal death in utero, intrapartum stillbirth, neonatal death, and death before hospital discharge of a liveborn infant.
Total duration of infant's first hospitalisation, in days | From date of infant birth to date of first discharge home from hospital (or date of death, whichever occurs earlier), assessed up to 12 months.
  Total duration of infant's first hospitalisation, in days. An average of three months.
Any breastmilk feeding (yes/no) at 42 weeks' postmenstrual age or day of first discharge home from hospital (whichever occurs earliest) | At 42 weeks' postmenstrual age or on day of first discharge home from hospital (whichever occurs earliest)
  Any breastmilk feeding at 42 weeks' postmenstrual age or on day of first hospital discharge home (whichever occurs earliest). Data will be collected as yes/no.
Number of infants with diagnosed patent ductus arteriosus (PDA) | At 42 weeks' postmenstrual age or on day of first discharge home from hospital (whichever occurs earliest)
  Number of infants diagnosed with PDA.
Number of infants diagnosed with retinopathy of prematurity (ROP) | At 42 weeks' postmenstrual age or on day of first discharge home from hospital (whichever occurs earliest)
  Number of infants diagnosed with retinopathy of prematurity (ROP). Worst stage and treatment will also be collected.
Number of infants who received postnatal corticosteroids | From date of trial entry to 42 weeks postmenstrual age or discharge home from hospital (whichever is earliest)
  Any postnatal corticosteroid and any mode of administration.
Maternal Outcome Set: Infant's birth weight z-score | At birth
  Infants birth weight z-score.
  This is a secondary outcome for Pregnancy Domains only.
Maternal Outcome Set: Infant's gestational age at birth | At birth
  Infant's gestational age at birth.
  This is a secondary outcome for Pregnancy Domains only.
Maternal Outcome Set: Number of maternal deaths | After trial entry and within 42 days postpartum
  Death of the mother or pregnant person.
  This is a secondary outcome for Pregnancy Domains only.
Maternal Outcome Set: Number of participants with severe maternal morbidity Maternal Outcome Set: Severe maternal morbidity | After trial entry and within 42 days postpartum
  Includes Intensive Care Unit (ICU) admission to an intensive care unit, sepsis, eclampsia, amniotic fluid embolism, pregnancy-related hysterectomy, severe primary postpartum haemorrhage, uterine rupture, cardiac arrest, endometritis, mechanical ventilation (not for birth), stroke).
  This is a secondary outcome for Pregnancy Domains only.
Maternal Outcome Set: Length of maternal hospitalisation, in days | From date of trial entry to date of discharge home from hospital (or date of death, whichever occurs earlier), assessed up to 12 months.
  Number of days from trial entry to hospital discharge, in days. An average of three weeks.
  This is a secondary outcome for Pregnancy Domains only.
Maternal Outcome Set: Number of participants readmitted to hospital | After trial entry AND after first discharge home from hospital AND within 42 days postpartum. Measured at 42 days postpartum, YES/NO and reason for re-admission.
  Readmission to hospital (any reason) after first hospital discharge and before 42 days postpartum.
  This is a secondary outcome for Pregnancy Domains only.
Maternal Outcome Set: Mode of birth | At birth
  Includes: vaginal birth, assisted vaginal birth, caesarean.
  This is a secondary outcome for Pregnancy Domains only.

CONTACTS AND LOCATIONS:
Overall Officials: Clare Whitehead, MBChB, PhD, Principal Investigator — University of Melbourne, Royal Women's Hospital, Melbourne.; Brett Manley, MBBS, PhD, Principal Investigator — University of Melbourne, Royal Women's Hospital, Melbourne

IPD SHARING:
Plan to Share IPD: Yes
Version 1, Apr-2024
  Once data unblinding no longer compromises the integrity of the trial, a de-identified data set collected for the analysis of domains within PLATIPUS will be made available.
  Conditions:
  1. All domains in which the participant is co-enrolled are closed to recruitment* (*Where one or more domains in which a participant is co-enrolled are not yet closed to recruitment, the participant's data may be provided, without the treatment code, to prevent unblinding in unfinished domains).
  2. Primary domain conclusions/analyses have been published, AND
  3. The 2-year follow-up of participants within the domain/s of interest is/are complete.
  Supporting materials (Core Protocol, Domain-Specific Appendices, Data Dictionaries and Domain-Specific Statistical Analysis Plans) will be available.
  Contact: University of Melbourne - info@platipustrial.org.
Supporting Information: Study Protocol, SAP
Time Frame: This is estimated to be approximately six months following the completion of the two-year follow-up of domain participants.
Access Criteria: To be determined. Access requests will be subject to review by trial subcommittees. The Trial Steering Committee will approve or disapprove requests. A Data Transfer Agreement and Authorship Agreement signed by relevant parties and evidence of ethical approval will be required.

REFERENCES:
- [Derived] Manley BJ, McKinlay CJD, Lee KJ, Groom KM, Whitehead CL. Adapt to survive and thrive: the time is now for adaptive platform trials for preterm birth. Lancet Child Adolesc Health. 2025 Feb;9(2):131-137. doi: 10.1016/S2352-4642(24)00328-6. PMID 39855752